CLINICAL TRIAL: NCT06743620
Title: Prospective Observational Long-Term Safety and Effectiveness Registry of Patients Who Have Received Iltamiocel as Part of Cook Myosite, Inc. Sponsored CELLEBRATE Clinical Study in Patients With Persistent or Recurrent Stress Urinary Incontinence (SUI) Following Surgical Treatment
Brief Title: Observational Registry for Iltamiocel Compared to Placebo for Urinary Sphincter Repair in Post-surgical Female Stress Incontinence
Acronym: CLBT RGST
Status: Enrolling by invitation | Type: Observational
Sponsor: Cook MyoSite (Industry)
Responsible Party: Sponsor
Other Study IDs: R15-06
Expanded Access: NCT04661293 (Available)
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with persistent or recurrent SUI following surgical treatment who have received iltamiocel
  Interventions: Other: iltamiocel

INTERVENTIONS:
Other: iltamiocel — This is an observational study with no intervention.

SUMMARY:
The main purpose of this registry is to collect observational, long-term safety and effectiveness data in subjects who have received at least one dose of iltamiocel as part of the CLBT clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Has completed participation within 15 months in the CLBT clinical study for females with persistent or recurrent SUI following surgical treatment (i.e., either subject has completed all follow-up visits or has been officially exited from the study).
* Has received at least one dose of iltamiocel as part of the CLBT study.
* Must be willing and able to comply with the study procedures, is able to understand all study requirements and must agree to read and sign the informed consent form prior to any study-related procedures.
* Has access to a phone or electronic device to allow completion of electronic documents

Exclusion Criteria:

* Has only received placebo as part of the CLBT study.
* Unable or unwilling to provide informed consent.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female subjects who have received iltamiocel as part of participation in the CLBT clinical study for females with persistent or recurrent SUI following surgical treatment will be considered for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2032-04 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Long term safety | 5 years
  Long term safety of iltamiocel
Long term effectiveness | 5 years
  Long term effectiveness of iltamiocel

CONTACTS AND LOCATIONS:
Overall Officials: Ron Jankowski, PhD, Study Director — Cook MyoSite, Inc.
Locations (1):
- Virtual Site, Harvard, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No